CLINICAL TRIAL: NCT01730573
Title: A Randomized Comparison of Inter Scalene and Combined Supra Scapular and Axillary Nerve Blocks for Postoperative Pain Relief in Arthroscopic Shoulder Rotator Cuff Repair
Brief Title: Interscalene and Combined Supra Scapular and Axillary Nerve Blocks in Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Professor, Department of Anaesthesia, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102994
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Disorder of Rotator Cuff
Keywords: interscalene; suprascapular; axillary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Active Comparator): This arm patients will receive inter scalene block which will be ultrasound and nerve stimulator guided.
  Interventions: Procedure: interscalene block
- Suprascapular and Axillary nerve block (Active Comparator): This arm patients will receive Suprascapular and axillary nerve blocks which will be ultrasound guided and nerve stimulator guided.
  Interventions: Procedure: Suprascapular and Axillary nerve block

INTERVENTIONS:
Procedure: interscalene block — This arm patients will receive inter scalene block which will be ultrasound and nerve stimulator guided.
  Arms: Interscalene block
Procedure: Suprascapular and Axillary nerve block — This arm patients will receive Suprascapular and axillary nerve blocks which will be ultrasound guided and nerve stimulator guided.
  Arms: Suprascapular and Axillary nerve block

SUMMARY:
Primary objective of this study is to prospectively compare and evaluate efficacy as well as note side effects of the interscalene block and combined suprascapular and axillary nerve block for ambulatory arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Patients having elective arthroscopic rotator cuff repair will be randomized to one of the two groups.

Group 1: This group will receive Interscalene block (ultrasound guided and nerve stimulator aided) followed by a general anesthesia.

Group 2: This group will receive Suprascapular and Axillary nerve block (ultrasound guided and nerve stimulator aided) followed by a general anesthesia.

Performance time, quality and efficacy as well as any side-effects of the blocks will be evaluated in terms of pain scores in recovery room, after 4- 6 hours and the next morning, opioid usage and patient satisfaction.

Primary hypothesis:

• Combined Suprascapular and axillary nerve blocks provide similar postoperative analgesia as compared to interscalene block for arthroscopic rotator cuff repair.

Secondary hypothesis

• Interscalene block is associated with more side effects and complications as compared to suprascapular nerve block and axillary nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Elective shoulder arthroscopic rotator cuff repair
* ASA I - III (American Society of Anaesthesia Classification)

Exclusion Criteria:

* ASA IV or higher ( American Society of Anaesthesia Classification)
* Obesity: BMI >35
* Narcotic Abuse/ Drug dependency
* Major Neurologic deficits
* Allergy to local anesthetics
* Infection in the site of the puncture
* Mental impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Analgesic Efficacy | one year
  Visual Analogue scores for pain will be analyzed using chi-squared test. Interscalene block (ISB) of the brachial plexus has been demonstrated to be one of the most effective analgesic modality during arthroscopic shoulder surgery. However, despite its (ISB) time-tested record of relative safety, ISB is associated with some complications. These could be central nervous system, respiratory and cardiovascular complications. These side effects and complications are based upon the anatomy of the brachial plexus at this level.Recently, suprascapular and axillary nerve blocks have been used to control postoperative shoulder pain. The study will try to find out whether combined supra scapular and axillary nerve blocks are as effective in pain control as compared to inter scalene block.

SECONDARY OUTCOMES:
Side effects | 1 year
  The study will try to find out whether combined supra scapular and axillary nerve blocks are associated with less side effects as compared to inter scalene block.

OTHER OUTCOMES:
Patient satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - St. Joseph's Health Care, London, Ontario
  - St. Joseph Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No